CLINICAL TRIAL: NCT07291102
Title: Comparison of Neurocognitive Outcome in Two Standard Regimen for Treatment of Low-risk Medulloblastoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: German Society of Paediatric Oncology and Hematology (GPOH gGmbH) (Unknown); Children's of Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COGNITO-MB; 2024-517133-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-21; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: "Head Start" 4 (Experimental): Arm A consists of 3 to 5 Induction chemotherapy cycles and one high-dose chemotherapy cycle evaluated in the "Head Start" 4 study.
  Interventions: Drug: Bridging Chemotherapy; Drug: Induction Cycles A1-A3; Drug: Induction Cycles A4-5; Drug: Consolidation Cycle A6
- Arm B: HIT-SKK (Experimental): Arm B consists of 3 to 5 cycles of chemotherapy evaluated in the HIT-SKK'92 (Rutkowski et al. 2005) and HIT-2000 (NCT00303810) clinical studies.
  Interventions: Drug: Bridging Chemotherapy; Drug: HIT-SKK Chemotherapy Cycles B1-3; Drug: Modified HIT-SKK Cycle B4-5

INTERVENTIONS:
Drug: Bridging Chemotherapy — One bridging chemotherapy cycle consists of five days of therapy using Carboplatin and etoposide
Drug: Induction Cycles A1-A3 — Cisplatin, vincristin, etoposide, cyclophosphamide, high-dose methotrexate
  Arms: Arm A: "Head Start" 4
Drug: Induction Cycles A4-5 — Cisplatin, etoposide, cyclophosphamide, high-dose methotrexate
  Arms: Arm A: "Head Start" 4
Drug: Consolidation Cycle A6 — Carboplatin, thiotepa, etoposide
  Arms: Arm A: "Head Start" 4
Drug: HIT-SKK Chemotherapy Cycles B1-3 — Cyclophosphamide, vincristine, high-dose methotrexate, carboplatin, etoposide, i.ventri. methotrexate
  Arms: Arm B: HIT-SKK
Drug: Modified HIT-SKK Cycle B4-5 — Cyclophosphamide, vincristine, carboplatin, etoposide
  Arms: Arm B: HIT-SKK

SUMMARY:
This is a trial to compare neurocognitive outcomes in the intent-to-treat population 2.5 years after diagnosis between patients with newly diagnosed, non-metastatic, SHH-activated, TP53-wt, non-MYC amplified MF randomized to the interventional arms A ("Head Start 4") or B (HIT-SKK).

DETAILED DESCRIPTION:
In this study, two highly effective irradiation-sparing treatment regimens are being compared in patients with low-risk early childhood MB:

1. Arm A: The "Head Start" 4 regimen developed by the North American Head Start Consortium. This approach uses intensive Induction chemotherapy and Consolidation with HDCT and has led to equally favorable results in this subgroup -- 3y PFS was 96% for infants and young children with M0, SHH MB; 5y EFS was 93% for M0, DMB on the predecessor "Head Start" 3 study.
2. Arm B: The HIT-SKK regimen developed within the GPOH. This regimen combines systemic chemotherapy with intraventricular MTX, leading to 93% 5-year PFS in low-risk patients.

Both treatment regimens use high-dose i.v. MTX, but only the HIT-SKK regimen also uses intraventricular administration of MTX directly into the CSF in addition to i.v. MTX. Given the long-term neurocognitive deficits of MTX have been described in childhood leukemia, and the pathogenesis of MTX-induced CNS-damage has been described, this has raised some concerns. Similarly, highly intensive, HDCT containing "Head Start" chemotherapy carries specific risks for the neurocognitive outcomes. Encouragingly, five years after HIT-SKK treatment including intraventricular MTX, young children with MB have a mean fluid intelligence score of 93.8 points. The full-scale IQ after "Head Start" chemotherapy is 95.4 and likewise within normal range. On the other hand, highly intensive, HDCT/AuHCR containing "Head Start" chemotherapy carries specific risks for the neurocognitive outcomes. However, neurocognitive outcomes after the HIT-SKK and "Head Start" chemotherapy regimens are difficult to compare from existing data, because of small sample sizes and inhomogeneous assessment tools used in prior studies. Therefore, a confirmatory study utilizing the same measures administered at the same time points is required to identify clinically relevant differences. In addition, survival, occurrence of second malignancies, neurological and endocrine deficits, hearing loss, and psychosocial comorbidities are also of high relevance in survivors of MB and may differ after both regimens. Since these also severely limit the survivors' potential for activity and participation in everyday life and affect their parents and siblings as well, this information will also be recorded.

ELIGIBILITY:
Inclusion Criteria for screening:

* Age at diagnosis < 5 years
* Patients with institutional suspicion or diagnosis of SHH-activated MB
* Patient and family in social circumstances that will allow neuropsychological follow-up
* Ability of parents/legal representatives to understand the patient information and to personally sign and date the informed consent to participate in screening procedures
* Patient and the parents/legal representative are able and willing to participate in the entire study (if patient is eligible)

Exclusion Criteria for overall study:

* Patients previously treated for any other brain tumor or any type of malignant disease
* Patients, in whom compliance with toxicity management guidelines and study procedures cannot be assured
* History of hypersensitivity to an investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of an investigational medicinal product.
* Patients/parents who do not wish to abstain from treatment with live vaccines during study participation
* Patients with a language barrier too extensive to complete neuropsychological tests based on the investigator's judgement
* Patients with severe premorbid developmental delay (based on the investigator's judgement), which will not allow WPPSI-IV assessment after 2.5 years
* Patients cannot undergo MRI

Inclusion Criteria for Bridging chemotherapy (carboplatin/etopiside) in interventional arms:

* Patients with SHH-activated MB, TP53-wt demonstrated by IHC for Gab1 or p75-NGFR, Yap1, beta-catenin, and TP53 (lack of strong and widespread nuclear p53 positivity) on central review according to WHO classification 2021.
* No clinical evidence of extra-CNS metastases
* Negative CSF cytology
* No prior therapy for MB other than surgery
* No other medical contraindications to chemotherapy:
* No uncontrolled invasive fungal infection or other severe systemic infection requiring system/parental therapy
* No other severe organ dysfunctions, which cannot be clinically controlled
* No concomitant use with yellow fever vaccine and with live virus and bacterial vaccines
* No demyelinating form of Charcot-Marie-Tooth syndrome
* Assessment of hearing function completed
* No evidence of cancer predisposition syndromes other than Gorlin syndrome or ELP1, GPR161 germline alterations.
* Provided written informed consent by parent(s)/parent representative(s) by bridging chemotherapy
* Patient should be enrolled within 28 days after diagnosis. Bridging chemotherapy can start as early as criteria for enrollment are met, and must start no later than 33 days after diagnosis

Exclusion Criteria for bridging chemotherapy:

* One or more of the inclusion criteria for bridging chemotherapy are lacking
* Other histology than SHH MB

Inclusion Criteria for randomization:

* Patient has received bridging chemotherapy as described in this protocol
* Patients with centrally reviewed SHH-activated MB, TP53-wt, according to WHO classification 2021
* Absence of metastatic disease on central radiology review
* Exclusion of TP53-mutation by DNA sequencing of the TP53-gene from tumor tissue by central review. Results from local institution will be accepted if raw data of this analysis is forwarded to the national central review institution
* Confirmation of SHH activation by DNA methylation-based classification on central review. Results from local institution will be accepted if raw data of this analysis is forwarded to the national central review institution
* No amplification of MYC (amplification of MYCN allowed). Array-based technologies (850k array, molecular inversion probe assay (MIP)), array-based comparative genomic hybridization (array-CGH) or next generation sequencing (NGS) DNA sequencing coverage MYC locus will be used. If these alternative assays give any indication of possible amplification, FISH will be performed on central review.
* No other medical contraindications to chemotherapy:
* No uncontrolled invasive fungal infection or other severe systemic infection requiring system/parental therapy
* No other severe organ dysfunctions, which cannot be clinically controlled
* No concomitant use with yellow fever vaccine and with live virus and bacterial vaccines
* No demyelinating form of Charcot-Marie-Tooth syndrome
* Retrospective assessment of pre-operative health-related QoL (HR-QoL) measured by Pediatric Quality of Life Inventory
* Provided written informed consent by parent(s)/parent representative(s) for randomization

Exclusion criteria for randomization:

-Patients are excluded from the interventional study if any of the following criteria are met:

1. One or more of the inclusion criteria for randomization are lacking
2. Patients with metastatic disease
3. TP53-mutated SHH MB
4. MYC amplified MB
5. Pre-existing condition incompatible with scheduled therapy (e.g. Fanconi anemia)
6. Patients with non-communicating hydrocephalus, e.g. due to perinatal intracranial haemorrhage, adueductal stenosis, or meningitis
7. Contraindication for any components of the randomized therapies, including HDCT and intraventricular chemotherapy. Note: postperative hydrocephalus is not a contraindication for i.ventr. MTX.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2034-10 (Estimated); Study Completion 2038-10 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Outcomes using WPPSIIV | 105 months
  To compare neurocognitive outcomes 2.5 years after diagnosis between patients randomized to the interventional arms A ("Head Start" 4) and B (HIT-SKK). Full-Scale Intelligence Quotient (IQ) as measured by the Wechsler Preschool and Primary Scale of Intelligence (WPPSIIV) administered to those between the ages of 2 years and 6 months to 7 years and 7 months old at 2.5 years after diagnosis (+/- 6 months).

SECONDARY OUTCOMES:
PFS | 152 months
  Progression-free survival (PFS) compared between randomized groups
rtPFS | 152 months
  Radiotherapy-free/progression-free survival (rtPFS) compared between randomized groups
OS | 152 months
  Overall survival (OS) compared between randomized groups
Second malignancies | 152 months
  Incidence of second malignancies compared between randomized groups
Number of patients with treatment-related adverse events as assessed by CTCAE v5.0 | 152 months
  Acute toxicities compared between randomized groups
Incidence of therapy-related deaths | 152 months
  Incidence of therapy-related deaths compared between randomized groups
Assessment of IQ in patients randomized to Head Start or HIT-SKK | 152 months
  Wechsler Intelligence Scale for Children (WISC-V) Full Scale IQ at 5 years after diagnosis (+/- 12 months range allowed), with the Wechsler Preschool and Primary Scale of Intelligence (WPPSI) Full Scale IQ Score used only for children < 6 years old.
Assessment of Development and Adaptive Functioning using ABAS v2 or v3 | 152 months
  Adaptive Behavior Assessment System (ABAS, versions II or 3) at diagnosis, 2.5- and 5 years after diagnosis will be used to compare patients randomized to Head Start or HIT-SKK.
Quality of Life Assessment using PedsQL Infant or PedsQL 4.0 parent-reported Quality of Life Measure | 152 months
  PedsQL Infant or PedsQL 4.0 parent-report QoL measure depending upon current age at the treatment timepoints. Questionnaires are quantified on a scale of 0-100 where higher scores indicate better outcomes/quality of life.
Correlation between neurocognitive outcomes and QoL | 152 months
  Correlation of neurocognitive outcomes (measured using WISC-V Full Scale IQ at 5 years after diagnosis) and quality of life (measured using PedsQL Infant) 5 years after diagnosis will be achieved using a regression for linear mixed model.
Assessment of impact on hearing using SIOP Boston scale | 152 months
  Ototoxicity will be assessed through hearing evaluation according to SIOP Boston scale (patients with normal Distortion-Product Otoacoustic Emissions (DPOAE) will be considered as not having hearing loss).
Number of patients with Leukoencephalopathy | 152 months
  LEP will be assessed 2.5 and 5 years after diagnosis compared between randomized groups using the modified Fazekas scale.
Compare PFS | 152 months
  To compare PFS between randomized groups in patients in CR at end of study therapy
Compare PFS | 152 months
  To compare PFS between subtypes of SHH-MB as defined by classification based on the Heidelberg brain tumor classifier Version 11 (or higher)
Assess rate of patients with cancer predisposition syndromes | 152 months
  To assess the rate of patients with genetically confirmed basal cell nevus syndrome (BCNS, Gorlin-Syndrome, OMIM: 109400), ELP1 and GPR161 cancer predisposition syndromes among eligible enrolled patients
Compare rtPFS | 152 months
  To compare rtPFS between subtypes of SHH-MB as defined by classification based on the Heidelberg brain tumor classifier Version 11 (or higher)
Compare OS | 152 months
  To compare OS between subtypes of SHH-MB as defined by classification based on the Heidelberg brain tumor classifier Version 11 (or higher)
Compare rtPFS | 152 months
  To compare rtPFS between randomized groups in patients in CR at end of study therapy
Compare OS | 152 months
  To compare OS between randomized groups in patients in CR at end of study therapy
Assessment of impact on hearing using Chang scales | 152 months
  Ototoxicity will be assessed through hearing evaluation according to Chang Scale (patients with normal Distortion-Product Otoacoustic Emissions (DPOAE) will be considered as not having hearing loss).
Association between neurocognitive and behavioral outcomes | 152 months
  Association of neurocognitive (measured using WISC-V Full Scale IQ at 5 years after diagnosis and WPPSI Full Scale IQ Score used only for children < 6 years old) outcomes and behavioral outcomes (measured using ABAS v2 or v3) 5 years after diagnosis compared between randomized groups

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, MD, Principal Investigator — Nationwide Children's Hospital; Girish Dhall, MD, Study Chair — Children's Hospital of Alabama
Locations (2):
- United States (2):
  - Children's of Alabama, Birmingham, Alabama
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
This study is considered for publication in the scientific literature in a peer re-viewed journal, irrespective of the results. Study results may also be presented at one or more medical congresses and may be used for scientific exchange and teaching purposes. Additionally, this study and its results may be submitted for inclusion in all appropriate health authority study registries, as well as publication on health authority study registry websites, as required by local health authority regulations.